CLINICAL TRIAL: NCT01061333
Title: A Two-Part, Randomized, Placebo-Controlled, Crossover Trial to Evaluate the Differential Effects of Inhaled Nedocromil, Oral Montelukast, and Inhaled Mometasone on Markers of the Early Airway Response to Allergen in Asthmatics
Brief Title: Early Airway Response to Allergen in Asthmatics (MK-0000-176)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-176; 2010_507 (Other: Merck)
Record Dates: First submitted 2010-02-01; First posted 2010-02-03 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Nedocromil; montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Experimental): Placebo
  Interventions: Drug: Placebo
- Montelukast (Experimental): Montelukast
  Interventions: Drug: Comparator: Montelukast
- Nedocromil (Experimental): Nedocromil
  Interventions: Drug: Nedocromil
- Mometasone (Experimental): Mometasone
  Interventions: Drug: Comparator: Mometasone

INTERVENTIONS:
Drug: Nedocromil — Nedocromil 4 mg, as metered dose inhaler 1 hour prior to allergen challenge
  Arms: Nedocromil
Drug: Comparator: Montelukast — Montelukast single 10 mg tablet administered 2 hours prior to allergen challenge
  Other Names: Singulair
  Arms: Montelukast
Drug: Comparator: Mometasone — Mometasone furoate 400 mcg by twisthaler, administered 2 hours prior to allergen challenge
  Arms: Mometasone
Drug: Placebo — Mometasone placebo twisthaler, Nedocromil placebo metered dose inhaler, Montelukast placebo tablet
  Arms: Placebo

SUMMARY:
This study will assess the Early Airway Response (EAR) associated change in forced expiratory volume in one second (FEV1) and plasma 9α-11ß-PGF2 ('9P') after single dose pretreatment of nedocromil, montelukast, and mometasone.

ELIGIBILITY:
Inclusion Criteria:

* History of mild to moderate Asthma
* In good general health (except for asthma)
* Stable and free of respiratory infection
* Nonsmoker
* Females highly unlikely to conceive (surgically sterilized, postmenopausal, or agrees to use 2 acceptable methods of birth control)

Exclusion Criteria:

* Nursing mother
* Recent or ongoing upper or lower respiratory tract infection
* Unable to refrain from or anticipates the use of any prescription and non-prescription drugs
* Consumes excessive amounts of alcohol or caffeine
* History of stroke, chronic seizures, or major neurological disorder
* History of cancer
* Received a vaccination within the past 3 weeks

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-06; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo-Montelukast-Nedocromil-Mometasone; Placebo-Nedocromil-Montelukast-Mometasone: Over the course of four 3-day treatment regimens, participants received a single dose of each drug starting with placebo, crossover of nedocromil or montelukast, crossover of nedocromil or montelukast, ending with mometasone; with a 20-day washout between each of the four treatment periods.
Period: Period 1: Placebo Run-in
Arm/Group | Placebo-Montelukast-Nedocromil-Mometasone | Placebo-Nedocromil-Montelukast-Mometasone
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Period 2: 20-day Washout
Arm/Group | Placebo-Montelukast-Nedocromil-Mometasone | Placebo-Nedocromil-Montelukast-Mometasone
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Period 3: Nedocromil-Montelukast X-over
Arm/Group | Placebo-Montelukast-Nedocromil-Mometasone | Placebo-Nedocromil-Montelukast-Mometasone
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Period 4: 20-day Washout
Arm/Group | Placebo-Montelukast-Nedocromil-Mometasone | Placebo-Nedocromil-Montelukast-Mometasone
Started | 8 | 8
Completed | 8 | 7
Not Completed | 0 | 1
Not completed — Discontinued by Study Team | 0 | 1
Period: Period 5: Nedocromil-Montelukast X-over
Arm/Group | Placebo-Montelukast-Nedocromil-Mometasone | Placebo-Nedocromil-Montelukast-Mometasone
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Period 6: 20-day Washout
Arm/Group | Placebo-Montelukast-Nedocromil-Mometasone | Placebo-Nedocromil-Montelukast-Mometasone
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Period 7: Mometasone
Arm/Group | Placebo-Montelukast-Nedocromil-Mometasone | Placebo-Nedocromil-Montelukast-Mometasone
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Over the course of four 3-day treatment regimens, participants received a single dose of each drug starting with placebo, nedocromil or montelukast, nedocromil or montelukast, ending with mometasone; with a 20-day washout between each of the four treatment periods.
Arm/Group | All Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.94 (7.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Forced Expiratory Volume in 1 Second (FEV1)
Description: Maximal percent drop in FEV1 at 20 minutes post allergen challenge
Time Frame: Pre-allergen challenge and 20 minutes after allergen challenge
Measure: Least Squares Mean (Standard Deviation); unit: Percentage drop in FEV1
Groups:
- Placebo: Nedocromil placebo metered dose inhaler, montelukast placebo tablet, mometasone placebo twisthaler
- Nedocromil: Nedocromil 4 mg, administered by metered dose inhaler, 1 hour prior to allergen challenge
- Montelukast: Montelukast 10 mg, administered in a single tablet, 2 hours prior to allergen challenge
- Mometasone: Mometasone furoate 400 mcg, administered by twisthaler, 2 hours prior to allergen challenge
Arm/Group | Placebo | Nedocromil | Montelukast | Mometasone
Number analyzed (Participants) | 16 | 16 | 15 | 15
Percentage drop in FEV1 | -24.66 (10.72) | -8.44 (6.15) | -9.15 (6.96) | -16.17 (11.01)
Statistical Analysis 1: Comparison: Placebo vs Nedocromil; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-value not adjusted for simultaneous multiple comparisons; Difference in LS mean = 16.22, 90% CI 2-sided [10.74 to 21.69]
Statistical Analysis 2: Comparison: Placebo vs Montelukast; Test type: Superiority or Other; p = 0.0001, ANCOVA — p-value not adjusted for simultaneous multiple comparisons; Difference in LS Mean = 15.51, 90% CI 2-sided [10.00 to 21.02]
Statistical Analysis 3: Comparison: Placebo vs Mometasone; Test type: Superiority or Other; p = 0.0432, ANCOVA — p-value not adjusted for simultaneous multiple comparisons; Difference in LS Mean = 8.49, 90% CI 2-sided [1.78 to 15.20]

2. Primary Outcome: Change in Plasma 9α-11β-PGF2 (9P) at 5 Minutes
Description: Fold change over baseline of plasma 9P at 5 minutes post-allergen challenge
Time Frame: Pre-allergen challenge and 5 minutes post allergen challenge
Measure: Geometric Mean (Standard Deviation); unit: Fold change over baseline
Arm/Group | Placebo | Nedocromil | Montelukast | Mometasone
Number analyzed (Participants) | 16 | 16 | 15 | 15
Fold change over baseline | 0.77 (0.21) | 0.97 (0.17) | 1.08 (0.44) | 1.00 (0.35)
Statistical Analysis 1: Comparison: Placebo vs Nedocromil; Test type: Superiority or Other; p = 0.0430, ANCOVA — p-Value not adjusted for simultaneous multiple comparisons; concentrations evaluated at log scale; Geom. Mean Ratio of fold over baseline = 1.27, 90% CI 2-sided [1.05 to 1.54]
Statistical Analysis 2: Comparison: Placebo vs Montelukast; Test type: Superiority or Other; p = 0.0100, ANCOVA — p-Value not adjusted for simultaneous multiple comparisons; concentrations evaluated at log scale; Geom. Mean Ratio of fold over baseline = 1.41, 90% CI 2-sided [1.15 to 1.72]
Statistical Analysis 3: Comparison: Placebo vs Mometasone; Test type: Superiority or Other; p = 0.0860, ANCOVA — p-Value not adjusted for simultaneous multiple comparisons; concentrations evaluated at log scale; Geom. Mean Ratio of fold over baseline = 1.30, 90% CI 2-sided [1.01 to 1.67]

3. Primary Outcome: Change in Plasma 9P at 20 Minutes
Description: Fold change over baseline of plasma 9P at 20 minutes post-allergen challenge
Time Frame: Pre-allergen challenge and 20 minutes post allergen challenge
Measure: Geometric Mean (Standard Deviation); unit: Fold change over baseline
Arm/Group | Placebo | Nedocromil | Montelukast | Mometasone
Number analyzed (Participants) | 16 | 16 | 15 | 15
Fold change over baseline | 1.22 (0.31) | 0.72 (0.25) | 0.72 (0.21) | 1.06 (0.40)
Statistical Analysis 1: Comparison: Placebo vs Nedocromil; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Value not adjusted for simultaneous multiple comparisons; concentrations evaluated at log scale; Geom. Mean Ratio of fold over baseline = 0.59, 90% CI 2-sided [0.50 to 0.70]
Statistical Analysis 2: Comparison: Placebo vs Montelukast; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Value not adjusted for simultaneous multiple comparisons; concentrations evaluated at log scale; Geom. Mean Ratio of fold over baseline = 0.59, 90% CI 2-sided [0.49 to 0.70]
Statistical Analysis 3: Comparison: Placebo vs Mometasone; Test type: Superiority or Other; p = 0.2679, ANCOVA — p-Value not adjusted for simultaneous multiple comparisons; concentrations evaluated at log scale; Geom. Mean Ratio of fold over baseline = 0.87, 90% CI 2-sided [0.69 to 1.08]

4. Secondary Outcome: Allergen-induced Changes in Urinary 9P
Description: Fold change over baseline in Urinary 9P at 2 hours post allergen challenge
Time Frame: Baseline and 2 hours post allergen challenge
Population: Only participants with baseline values were analyzed
Measure: Geometric Mean (Standard Deviation); unit: Fold change over baseline
Arm/Group | Placebo | Nedocromil | Montelukast | Mometasone
Number analyzed (Participants) | 13 | 14 | 14 | 13
Fold change over baseline | 1.54 (2.43) | 1.39 (2.54) | 1.45 (4.22) | 1.40 (2.24)
Statistical Analysis 1: Comparison: Placebo vs Nedocromil; Test type: Superiority or Other; p = 0.7622, ANCOVA — p-Value not adjusted for simultaneous multiple comparisons; concentrations evaluated at log scale; Geom. Mean Ratio of fold over baseline = 0.90, 90% CI 2-sided [0.51 to 1.59]
Statistical Analysis 2: Comparison: Placebo vs Montelukast; Test type: Superiority or Other; p = 0.8468, ANCOVA — p-Value not adjusted for simultaneous multiple comparisons; concentrations evaluated on log scale; Geom. Mean Ratio of fold over baseline = 0.94, 90% CI 2-sided [0.53 to 1.65]
Statistical Analysis 3: Comparison: Placebo vs Mometasone; Test type: Superiority or Other; p = 0.6140, ANCOVA — p-Value not adjusted for simultaneous multiple comparisons; concentrations evaluated at log scale; Geom. Mean Ratio of fold over baseline = 0.91, 90% CI 2-sided [0.65 to 1.26]

5. Secondary Outcome: Allergen-induced Changes in Urinary Leukotriene (LT) E4
Description: Fold change over baseline in urinary LTE4 at 2 hours post-allergen challenge
Time Frame: Baseline and 2 hours post allergen challenge
Population: Only participants with baseline values were analyzed
Measure: Geometric Mean (Standard Deviation); unit: Fold change over baseline
Arm/Group | Placebo | Nedocromil | Montelukast | Mometasone
Number analyzed (Participants) | 13 | 14 | 14 | 13
Fold change over baseline | 1.77 (1.09) | 1.19 (1.31) | 1.40 (1.52) | 1.62 (1.35)
Statistical Analysis 1: Comparison: Placebo vs Nedocromil; Test type: Superiority or Other; p = 0.0006, ANCOVA — p-Value not adjusted for simultaneous multiple comparisons; concentrations evaluated at log scale; Geom. Mean Ratio of fold over baseline = 0.67, 90% CI 2-sided [0.57 to 0.80]
Statistical Analysis 2: Comparison: Placebo vs Montelukast; Test type: Superiority or Other; p = 0.0291, ANCOVA — p-Value not adjusted for simultaneous multiple comparisons; concentrations evaluated at log scale; Geom. Mean Ratio of fold over baseline = 0.79, 90% CI 2-sided [0.67 to 0.94]
Statistical Analysis 3: Comparison: Placebo vs Mometasone; Test type: Superiority or Other; p = 0.3738, ANCOVA — p-Value not adjusted for simultaneous multiple comparisons; concentrations evaluated at log scale; Geom. Mean Ratio of fold over baseline = 0.92, 90% CI 2-sided [0.77 to 1.08]

6. Secondary Outcome: Allergen-induced Concentrations of Sputum LTC4
Description: Concentrations of LTC4 in sputum at 2 hours post-allergen challenge
Time Frame: 2 hours post allergen challenge
Population: Pre-imputation status. Missing data points were excluded and values below the lower limit of quantification (LLOQ) were included in the analysis with an assigned value of assay LLOQ.
Measure: Geometric Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Nedocromil | Montelukast | Mometasone
Number analyzed (Participants) | 16 | 16 | 14 | 14
pg/mL | 13.63 (8.22) | 14.02 (12.53) | 13.76 (5.45) | 12.14 (6.94)
Statistical Analysis 1: Comparison: Placebo vs Nedocromil; Test type: Superiority or Other; p = 0.7501, ANOVA — p-Value not adjusted for simultaneous multiple comparisons; concentrations evaluated at log scale; Geom. mean of fold change over Placebo = 1.03, 90% CI [0.88 to 1.20]
Statistical Analysis 2: Comparison: Placebo vs Montelukast; Test type: Superiority or Other; p = 0.9410, ANOVA — p-Value not adjusted for simultaneous multiple comparisons; concentrations evaluated at log scale; Geom. mean of fold change over Placebo = 1.01, 90% CI 2-sided [0.81 to 1.25]
Statistical Analysis 3: Comparison: Placebo vs Mometasone; Test type: Superiority or Other; p = 0.1165, ANOVA — p-Value not adjusted for simultaneous multiple comparisons; concentrations evaluated at log scale; Geom. mean of fold change over Placebo = 0.89, 90% CI 2-sided [0.79 to 1.01]

7. Secondary Outcome: Allergen-induced Concentrations of Sputum LTD4
Description: Concentrations of LTD4 in sputum at 2 hours post-allergen challenge
Time Frame: 2 hours post allergen challenge
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Nedocromil | Montelukast | Mometasone
Number analyzed (Participants) | 16 | 16 | 14 | 14
pg/mL | 17.48 (15.20) | 18.04 (31.13) | 18.52 (9.22) | 17.37 (36.91)
Statistical Analysis 1: Comparison: Placebo vs Nedocromil; Test type: Superiority or Other; p = 0.8616, ANOVA — p-Value not adjusted for simultaneous multiple comparisons; concentrations evaluated at log scale; Geom. mean of fold change over Placebo = 1.03, 90% CI 2-sided [0.76 to 1.41]
Statistical Analysis 2: Comparison: Placebo vs Montelukast; Test type: Superiority or Other; p = 0.7512, ANOVA — p-Value not adjusted for simultaneous multiple comparisons; concentrations evaluated at log scale; Geom. mean of fold change over Placebo = 1.06, 90% CI 2-sided [0.77 to 1.45]
Statistical Analysis 3: Comparison: Placebo vs Mometasone; Test type: Superiority or Other; p = 0.9723, ANOVA — p-Value not adjusted for simultaneous multiple comparisons; concentrations evaluated at log scale; Geom. mean of fold change over Placebo = 0.99, 90% CI 2-sided [0.72 to 1.37]

8. Secondary Outcome: Allergen-induced Concentrations of Sputum LTE4
Description: Concentrations of LTE4 in sputum at 2 hours post-allergen challenge
Time Frame: 2 hours post allergen challenge
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Nedocromil | Montelukast | Mometasone
Number analyzed (Participants) | 16 | 16 | 14 | 14
pg/mL | 115.5 (129.0) | 149.8 (178.7) | 181.3 (227.6) | 140.3 (215.8)
Statistical Analysis 1: Comparison: Placebo vs Nedocromil; Test type: Superiority or Other; p = 0.1983, ANOVA — p-Value not adjusted for simultaneous multiple comparisons; concentrations evaluated at log scale; Geom. mean of fold change over Placebo = 1.30, 90% CI 2-sided [0.92 to 1.82]
Statistical Analysis 2: Comparison: Placebo vs Montelukast; Test type: Superiority or Other; p = 0.0872, ANOVA — p-Value not adjusted for simultaneous multiple comparisons; concentrations evaluated at log scale; Geom. mean of fold change over Placebo = 1.57, 90% CI 2-sided [1.02 to 2.42]
Statistical Analysis 3: Comparison: Placebo vs Mometasone; Test type: Superiority or Other; p = 0.2499, ANOVA — p-Value not adjusted for simultaneous multiple comparisons; concentrations evaluated at log scale; Geom. mean of fold change over Placebo = 1.22, 90% CI 2-sided [0.91 to 1.62]

ADVERSE EVENTS:
Arm/Group | Placebo | Nedocromil | Montelukast | Mometasone
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 5/16 | 4/16 | 3/15 | 0/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | Nedocromil (N=16) | Montelukast (N=15) | Mometasone (N=15)
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Influenza Like Illness (General disorders) | 1 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0
Joint Sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 2 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For multicenter studies, subsequent to the multicenter publication, an investigator and colleagues may publish their data independently. Limitations of single site observations should always be described in such a manuscript. The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 60 days prior to submission. Any information identified by the SPONSOR as confidential must be deleted prior to submission.